CLINICAL TRIAL: NCT02622854
Title: Comparison of Plasma Exchange and Conservative Management in Non-severe Acute Hypertriglyceridemic Pancreatitis With Mildly Elevated Triglycerides
Brief Title: Plasma Exchange vs Conservative Management in Non-severe Acute Hypertriglyceridemic Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Jakob Gubensek, MD, PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HiperlipPankr
Record Dates: First submitted 2015-11-26; First posted 2015-12-07 (Estimated); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Acute Pancreatitis
Keywords: plasma exchange; hypertriglyceridemia
MeSH Terms: conditions — Pancreatitis; Hypertriglyceridemia | interventions — Plasma Exchange; Conservative Treatment; Glucose; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- plasma exchange (Experimental): plasma exchange, with 1.5 estimated plasma volume exchanged with albumin solution, using citrate anticoagulation, performed daily until triglycerides <=10 mmol/l
  Interventions: Procedure: plasma exchange
- conservative treatment (Active Comparator): infusion of 5% glucose and insulin, to maintain blood glucose at 5-8 mmol/l
  Interventions: Drug: conservative treatment

INTERVENTIONS:
Procedure: plasma exchange — see arm description
  Arms: plasma exchange
Drug: conservative treatment — see arm description
  Other Names: glucose and insulin
  Arms: conservative treatment

SUMMARY:
To compare effectiveness in reducing triglycerides between daily plasma exchange and glucose+insulin infusion in patients with non-severe acute hypertriglyceridemic pancreatitis with mildly elevated triglycerides

ELIGIBILITY:
Inclusion Criteria:

* mild acute hypertriglyceridemic pancreatitis
* triglycerides >15 but < 40 mmol/l

Exclusion Criteria:

* pregnancy
* severe course of pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-06; Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
decrease in triglycerides | within first 24 h after admission
  as % of starting value

SECONDARY OUTCOMES:
time until triglycerides drop to <10 mmol/l | by the end of hospital stay, up to 100 days
  expressed in days
highest C-reactive protein (CRP) | by the end of hospital stay, up to 100 days
% of patients with severe pancreatitis | by the end of hospital stay, up to 100 days

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Gubensek, MD, PhD, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia, Ljubljana, Slovenia

REFERENCES:
- [Result] Gubensek J, Andonova M, Jerman A, Persic V, Vajdic-Trampuz B, Zupunski-Cede A, Sever N, Plut S. Comparable Triglyceride Reduction With Plasma Exchange and Insulin in Acute Pancreatitis - A Randomized Trial. Front Med (Lausanne). 2022 Apr 12;9:870067. doi: 10.3389/fmed.2022.870067. eCollection 2022. PMID 35492338